CLINICAL TRIAL: NCT05344508
Title: Brensocatib in Patients With Non-Cystic Fibrosis Bronchiectasis
Brief Title: An Expanded Access Study to Assess Brensocatib for Participants With Non-Cystic Fibrosis Bronchiectasis
Status: Approved for marketing | Type: Expanded Access
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: INS1007-EAP
Record Dates: First submitted 2022-04-06; First posted 2022-04-25 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Non-Cystic Fibrosis Bronchiectasis
Keywords: Cathepsin G; CKD-EPI; NCFBE
MeSH Terms: interventions — brensocatib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Brensocatib — Brensocatib tablets

SUMMARY:
The purpose of this study is to allow early access to brensocatib for participants with non-cystic fibrosis bronchiectasis (NCFBE) who have successfully completed the INS1007301 ASPEN Clinical trial.

DETAILED DESCRIPTION:
Participants will receive brensocatib 10 mg, oral tablets, once daily.

ELIGIBILITY:
Inclusion Criteria:

* Participant had agreed to provide their informed consent to participate per local requirements.
* Participant had successfully completed Clinical Trial INS 1007-301 ASPEN, including the End of study Visit 12 prior to receiving treatment.
* Requests for Post-Trial access for brensocatib had come from ASPEN investigator.
* Had received brensocatib treatment.

Exclusion Criteria:

* Participant had experienced a serious adverse event deemed to be related to brensocatib during the study and required permanent participant is continuation.
* The participant is immunocompromised or chronically treated with any investigational or commercialized immunomodulatory agent that is directed to any component of the adaptive or innate immune systems.

Note: The use of any immunomodulatory agents (including but not limited to: bortezomib, ixazomib, thalidomide, cyclophosphamide, mycophenolate, Janus kinase inhibitors, IFN-γ, and azathioprine) is prohibited during the program.

* The participant had undergone continuous use of high dose non-steroidal anti-inflammatory drugs.
* The participant had undergone chronic use of systemic steroids for any chronic condition, except steroids with topical anti-inflammatory activities (ie, oral budesonide).
* Participant had planned to receive live attenuated vaccines during the program (treatment must be postponed until 4 weeks after the last dose of drug).
* Participant had planned to use investigational drugs.

Ages: 12 Years to 85 Years | Sex: All
Age Groups: Child, Adult, Older Adult